CLINICAL TRIAL: NCT03657615
Title: Hearing Aid Impact on Chronic Tinnitus Patients With Associated Hearing Loss Evaluated by Resting State Positron Emission Tomography (PET).
Brief Title: Hearing Aid Impact on Chronic Tinnitus Patients Evaluated by Resting State PET.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USaoPauloCF
Record Dates: First submitted 2018-07-11; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-07

CONDITIONS: Chronic Tinnitus
Keywords: hearing loss; tinnitus; neuroimaging; hearing aids; Positron emission Tomography - PET
MeSH Terms: conditions — Hearing Loss; Tinnitus

STUDY DESIGN:
Intervention Model Description: within subject
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Hearing Aid Fitting Patients with hearing loss but no tinnitus paired by age and hearing loss degree Hearing aided fitted PET image acquisition before and after 6 months og Hearing aid usage.
  Interventions: Device: hearing aid fitting
- Tinnitus (Experimental): Hearing Aid Fitting Patients with tinnitus and hearing loss associated Hearing aided fitted PET image acquisition before and after 6 months og Hearing aid usage.
  Interventions: Device: hearing aid fitting

INTERVENTIONS:
Device: hearing aid fitting — All patients were fitted bilaterally with hearing aids for hearing loss compensation. . Apart from different HAs used, device selection followed strict criteria to fit hearing loss demands, patient profile, resources and algorithms recommended for tinnitus patients.
  Other Names: hearing amplification

SUMMARY:
Using resting state positron emission tomography (PET), our goal was to analyze the metabolic and functional neural changes that occur after 6 months of effective hearing aid (HA) use. Besides, we correlate those changes with behavioral results. Patients with chronic tinnitus and untreated sensorineural hearing loss were tested pre-HA fitting, and at 6 months post-HA fitting.

DETAILED DESCRIPTION:
Subjects are selected as they are enrolled in the Tinnitus Research Group between January 2014 and September 2018. The study was approved by the local medical ethics committee for research at the Medical School of University of São Paulo - protocol number 611.174 in April, 2014.

All the procedures were performed after medical evaluation and a complete tinnitus evaluation protocol, which included somatosensory assessment, self-related questionnaires for tinnitus and hearing: Tinnitus Handicap Inventory (THI), Hearing Handicap Inventory for Adults (HHIA), and , for anxiety and depression symptoms: Generalized Anxiety Depression Scale (GAD-7) and Patient Health Questionnaire (PHQ-9), and for neck pain (Neck Disability Index, NDI). The subjects of this study were also blood tested for pregnancy and diabetes, which may interfere on fluorodeoxyglucose (FDG)-positron emission tomography PET acquisition.

All subjects underwent hearing and tinnitus evaluation, counseling and hearing aid fitting.

To prescribe and verify acoustic response, we used the HA fitting protocol recommended by the National Acoustics Laboratories (NAL), named NAL NL-2 (NL-non linear) FDG-PET measurements were obtained at baseline (prior to HA fitting) and after 6 months of HA use.

Regarding FDG-PET images, a within-subject analysis was performed by comparing pre-treatment and post-treatment group using paired-t-tests.

ELIGIBILITY:
Inclusion Criteria::

1. chronic perception of tinnitus for more than 6 months;
2. THI score greater than 38;
3. bilateral and symmetric hearing loss not exceeding 70 decibels (dB) hearing threshold;
4. no previous experience with HA. -

Exclusion Criteria:

1. unilateral, mixed or conductive hearing loss;
2. pulsatile or myoclonic tinnitus;;
3. anxiety and depression detected by GAD-7 and PHQ-9;
4. significant visual, motor or cognitive deficits;
5. pregnant women and diabetic patients
6. history of drug abuse -

Ages: 32 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01-15 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
PET RESULTS | 6 months
  After an individual whole brain analysis, a within-subject analysis was performed by comparing pre-treatment and post-treatment situation. The analysis revealed increased and decreased glycolytic metabolism areas for each subject, after intervention. For group analysis we used paired-t-tests. These analyses produced parametric statistical maps, which were then converted into a normal distribution unit (Z-scores). The significance threshold was set at p<0.05, and corrected for multiple comparisons (FWE or family-wise error rate), either at the voxel or cluster-level.

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 6 months
  The THI consists of 25 questions distributed on three scales that evaluate different tinnitus aspects: functional, emotional and catastrophic. The options for responding to THI questions are: yes (4 points), sometimes (2 points), and no (0 points). On a scale from 0-100, 0-16 points signifies negligible tinnitus, 18-36 signifies mild tinnitus, 38-56 signifies moderate tinnitus, 58-76 signifies severe tinnitus, and 78-100 signifies catastrophic tinnitus. Reductions on scale signifies tinnitus perception are reduced.Results of self-assessment questionnaires and their respective subscales were described according to the follow up evaluation moment. They were all analyzed statistically.
Hearing Handicap Inventory for Adults (HHIA) | 6 months
  Composed of 25 questions that evaluate social and emotional aspects of hearing disability. Subjects had three choices: yes (4 points), sometimes (2 points) and no (0 points). On a scale from zero to 100, scores higher than 44 points indicate severe handicap, from 18-42 points indicate moderate handicap and below 18 indicate no handicap. After intervention, reductions on scale means less hearing handicap.Results of self-assessment questionnaires and their respective subscales were described according to the follow up evaluation moment. They were all analyzed statistically.
Visual Analog Scale ( VAS) | 6 months
  The VAS is a numeric scale ranging from 0-10. Subjects assigned a value to tinnitus annoyance based on this visual scale. High scores means high degree of tinnitus annoyance.Results were described according to the follow up evaluation moment. and then analyzed statistically.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No